CLINICAL TRIAL: NCT06656416
Title: A Randomized, Double-Blind, Placebo-Controlled Study Followed by Open-Label Treatment of ALTO-100 in Adults With Bipolar Disorder Currently Experiencing a Major Depressive Episode
Brief Title: ALTO-100 in Bipolar Disorder With Depression (BD-D)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTO-100-211
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Disorder I or II With a Major Depressive Episode
Keywords: Bipolar I; Bipolar II; Major Depressive Episode

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALTO-100 (Experimental): Participants will receive ALTO-100 40 mg tablet twice daily, from Day 1 to Week 6 in the double blind (DB) treatment period. Eligible participants who enter the open label (OL) treatment period will receive ALTO-100 40 mg tablet twice daily from OL baseline until the end of OL period/early termination visit (Up to 7 weeks).
  Interventions: Drug: ALTO-100
- Placebo DB (Placebo Comparator): Participants will receive matching placebo tablet twice daily, from Day 1 to Week 6 in the double blind (DB) treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALTO-100 — ALTO-100 40 mg tablet BID
  Arms: ALTO-100
Drug: Placebo — Placebo tablet BID
  Arms: Placebo DB

SUMMARY:
The purpose of this study is to assess antidepressant efficacy differences between ALTO-100 and placebo during the Double-Blind period in patients with bipolar disorder I or II with current major depressive episode, when used adjunctively to a mood stabilizer and/or atypical antipsychotic, related to patient characteristics. Additionally, safety, tolerability, and efficacy will be assessed in a subsequent open label treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of BD-I or BD-II as well as BD-D
* At baseline, taking a mood stabilizer, lithium (LI) or lamotrigine (LMG) or valproic acid (VPA, any form) or combination of Li + LMG or Li + VPA and/or taking an approved atypical antipsychotic medication (olanzapine, quetiapine, lurasidone, risperidone, ziprasidone, cariprazine, aripiprazole, lumateperone, and asenapine) for at least 6 weeks with no dose modifications in the past 2 weeks
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study

Exclusion Criteria:

* Evidence of unstable medical condition
* Concurrent use of any prohibited medications or substance use disorder
* Diagnosed psychotic disorder (other than mania or depression)
* Current moderate or severe substance use disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-100 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess efficacy of ALTO-100 versus placebo on depression symptoms in bipolar disorder in a pre-defined subgroup of participants as measured by the mean change from Day 1 to Week 6 on the Montgomery-Åsberg Depression Rating Scale (MADRS) total score | Change assessed from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
To assess efficacy of ALTO-100 vs placebo for self-reported depressive symptoms in bipolar disorder patients in a pre- defined subgroup of participants as measured by the change from Day 1 to Week 6 in Patient Health Questionnaire, 9 item (PHQ-9) | Assessed 4 times over a 6-week interval, from Day 1 to Week 6
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders-5th edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4- point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
To assess efficacy of ALTO-100 vs placebo in severity of bipolar disorder symptoms in a pre-defined subgroup of participants as measured by the change from Day 1 to Week 6 in Clinician Global Impression Scale-severity (CGI-S) | Assessed 4 times over a 6-week interval, from Day 1 to Week 6
  The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of illness exhibited by a participant, rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill;5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 vs placebo for depressive symptoms in MDD in a pre-defined subgroup as measured by the change from Day 1 to Week 6 in response (>50% improvement from baseline) and remission (total score of <10) rates based on MADRS | Assessed 4 times over a 6-week interval, from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 vs placebo on depressive symptoms in bipolar disorder in all randomized participants as measured by the change from Day 1 to Week 6 on the MADRS | Assessed 4 times over a 6-week interval, from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To evaluate the safety of ALTO-100 during both the DB and OL periods of the study as measured by the assessment of the incidence, severity, and relatedness of Treatment Emergent Adverse Events (TEAEs), SAEs, discontinuation due to TEAEs and deaths | Assessed from Day 1 to Week 13
To evaluate the safety of ALTO-100 during both the DB and OL periods of the study as measured by the assessment of Heart Rate in bpm | Assessed from Day 1 to Week 13
  Assessment of Heart Rate in bpm
To evaluate the safety of ALTO-100 during both the DB and OL periods of the study as measured by the assessment of Blood Pressure in mmHg | Assessed from Day 1 to Week 13
  Assessment of Blood Pressure in mmHg
To evaluate the safety of ALTO-100 during both the DB and OL periods of the study as measured by the assessment of Weight in pounds | Assessed from Day 1 to Week 13
  Assessment of Weight in pounds
To evaluate the safety of ALTO-100 during both the DB and OL periods of the study as measured by the assessment of suicidality with the Concise Health Risk Tracking Self-Report,12 item scale (CHRT-SR12) | Assessed from Day 1 to Week 13
  The CHRT is a brief, self-report measure that systematically assesses both suicidal thinking and associated thoughts that may indicate the propensity for suicidal acts. The CHRT-SR12 is a 12 item scale. The patient assigns a score of 0-4for each item of the scale, allowing for a total score of 0 to 48, with the higher score signifying more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Savitz, MD, PhD, Study Director — Alto Neuroscience
Locations (27):
- United States (27):
  - Site 6036, Chandler, Arizona
  - Site 6000, Phoenix, Arizona
  - Site 6087, Yuma, Arizona
  - 6039, Fayetteville, Arkansas
  - 6070, Little Rock, Arkansas
  - Site 6081, Imperial, California
  - 6069, Los Angeles, California
  - Site 6016, Mather, California
  - Site 6082, Oceanside, California
  - Site 6102, Riverside, California
  - Site 6112, Colorado Springs, Colorado
  - Site 6067, Lauderhill, Florida
  - Site 6068, Atlanta, Georgia
  - Site 6064, Peachtree Corners, Georgia
  - Site 6151, Baltimore, Maryland
  - Site 6076, Bel Air, Maryland
  - Site 6062, Gaithersburg, Maryland
  - Site 6142, Lincoln, Nebraska
  - Site 6144, Las Vegas, Nevada
  - Site 6104, Las Vegas, Nevada
  - Site 6066, Toms River, New Jersey
  - Site 6014, Albuquerque, New Mexico
  - Site 6078, Albuquerque, New Mexico
  - 6065, North Canton, Ohio
  - Site 6075, Westlake, Ohio
  - Site 6072, Houston, Texas
  - Site 6121, Draper, Utah

IPD SHARING:
Plan to Share IPD: No